CLINICAL TRIAL: NCT06372457
Title: mavaCamten ObservationaL evIdence Global cOnsortium in HCM (COLLIGO-HCM)
Brief Title: COLLIGO-HCM: A Multinational Observational Study of the Real-World Effectiveness of Mavacamten Among Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy (oHCM)
Acronym: COLLIGO-HCM
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1107
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: mavacamten, oHCM, cardiac myosin inhibitor, NYHA class, echocardiogram parameters, patient-reported outcomes
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Hypertrophic Cardiomyopathy (HCM): Participants with an available HCM diagnosis date and without evidence of an HCM phenocopy
  Interventions: Drug: Approved Hypertrophic Cardiomyopathy drug treatments
- Participants treated with mavacamten.
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Approved Hypertrophic Cardiomyopathy drug treatments — As per product label
  Groups: Participants with Hypertrophic Cardiomyopathy (HCM)
Drug: Mavacamten — As per product label
  Groups: Participants treated with mavacamten.

SUMMARY:
COLLIGO-HCM is a global observational study that will conduct observational research of hypertrophic cardiomyopathy (HCM) treatment in real-world clinical practice.

DETAILED DESCRIPTION:
The mavaCamten ObservationaL evIdence Global cOnsortium in hypertrophic cardiomyopathy (COLLIGO-HCM) is a global observational research initiative aiming to describe the real-world outcomes of treatments for obstructive hypertrophic cardiomyopathy (HCM), including mavacamten.

This retrospective study uses data from existing medical records and electronic registries from HCM centers around the world.

ELIGIBILITY:
Inclusion Criteria:

* Source Cohort

  - Have at least one recorded encounter with a Hypertrophic Cardiomyopathy (HCM) diagnosis during or after 2018 (the first is defined as the index) and aged ≥18 years on the index date.

  - Disease-specific patient history documented in the medical record.
* HCM Sub-Cohort

  - Participants in the source cohort with a known HCM diagnosis
* Mavacamten Sub-Cohort - Participants who have their first mavacamten prescription after the index date

Exclusion Criteria:

• HCM Sub-Cohort

- HCM phenocopy (athlete's heart, hypertensive heart disease, Fabry disease, Pompe disease, Danon disease, amyloidosis) observed after the first observed HCM-associated encounter in the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients who have been diagnosed with Hypertrophic Cardiomyopathy (HCM).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Participant age at Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline, index date
Participant age at mavacamten treatment initiation | Index date
Participant sex | Baseline
Participant race/ethnicity | Baseline
Participant insurance coverage | Baseline
Participant employment status | Baseline
Participant educational level | Baseline
Date of Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline or index date
Participant body mass index (BMI) at Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline or index date
Hypertrophic Cardiomyopathy (HCM) subtype at diagnosis | Baseline or index date
Participant echocardiogram (ECHO) parameters at Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline or index date, and up to 33 months
Participant New York Heart Association (NYHA) class | Baseline or index date, and up to 33 months
Reason/trigger for initiating the path to Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline
Date of reason/trigger that initiated the path to Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline
Participant height | Baseline
Participant weight | Baseline
Participant blood pressure | Baseline
Participant heart rate | Baseline
Participant Hypertrophic Cardiomyopathy (HCM) symptoms | Baseline or index date, and up to 33 months
European participant CYP2C19 genotype | Baseline or index date, and up to 33 months
Participant family history of Hypertrophic Cardiomyopathy (HCM) | Baseline or index date
Participant family history of obstructive Hypertrophic Cardiomyopathy o(HCM) | Baseline or index date
Participant family history of sudden cardiac death (SCD) | Baseline or index date
Participant smoking status | Baseline or index date
Participant alcohol use | Baseline or index date
Participant recreational drug use | Baseline or index date
Participant involvement in a Hypertrophy Cardiomyopathy (HCM) randomized clinical trial (RCT) | Baseline or index date, and up to 33 months
Participant cardiovascular (CV) and CV-related comorbidities | Baseline and index date
  Comorbidities include:
  * Aortic stenosis
  * Cardiomyopathies, other (dilated, restrictive, arrhythmogenic right ventricular dysplasia, takotsubo cardiomyopathy)
  * Chronic kidney disease
  * Coronary heart disease
  * Deep venous thrombosis (DVT)
  * Heart failure
  * Hyperlipidemia
  * Hypertension
  * Hypertensive renal disease
  * Mitral valve prolapse
  * Peripheral vascular disease
  * Pulmonary hypertension
  * Phenocopy disorders (athlete's heart, hypertensive heart disease, Fabry disease, Pompe disease, Danon disease, amyloidosis)
Participant non-cardiovascular (CV)-related comorbidities | Baseline or index date
  Including:
  * Anxiety/panic attacks
  * Asthma
  * COPD
  * Depression
  * Diabetes
  * Liver diseases
Participant electrocardiogram (ECG) rhythm results | Baseline or index date
Participant cardiac magnetic resonance imaging (MRI) results | Baseline or index date
Participant N-terminal pro-B-type natriuretic peptide (NT-proBNP) results | Baseline or index date
Participant cardiac troponin results | Baseline or index date
Participant cardiopulmonary exercise test (CPET) results | Baseline or index date
Participant cardiac monitoring results | Baseline or index date
Participant exercise test results | Baseline or index date
Participant blood creatine levels | Baseline or index date
Participant cardiovascular (CV) events | Baseline
  Cardiovascular events include:
  * Atrial fibrillation
  * Atrial flutter
  * Myocardial infarction (MI)
  * Stroke
  * Transient ischemic attack (TIA)
  * Cardiac arrest
  * Sudden cardiac death (SCD)
  * Arrhythmia
  * Heart failure exacerbation
  * Incident heart failure
  * Ventricular fibrillation
  * Syncope
Type of procedures received by participants | Baseline or index date, and up to 33 months
  Procedures include:
  * Septal reduction therapy (SRT)
  * Implantable cardioverter defibrillator (ICD), including CRT-D
  * Pacemaker
  * Cardiac resynchronization therapy (CRT)
  * Atrial fibrillation ablation
  * Cardioversion
  * Heart transplant/use of ventricular assist device
  * Heart failure monitoring (e.g., CardioMEMS)
  * Percutaneous cutaneous intervention (PCI)
Cardiovascular treatments prescribed to participants | Baseline, and up to 33 months
Date of mavacamten prescription | Baseline
Date of mavacamten treatment initiation | Index date
Date of mavacamten dosage change | Up to 33 months
Reason for mavacamten dosage change | Up to 33 months
Occurrence of mavacamten stable dose (a period of 6-months with the same dose) | Up to 33 months
Dates of follow-up after mavacamten treatment initiation | Up to 33 months
Date of mavacamten treatment interuption or discontinuation | Up to 33 months
Reason for mavacamten treatment interuption or discontinuation | Up to 33 months
Supportive care provided to participants | Up to 33 months
Heath care resource utilization (HCRU) | Up to 33 months
Hypertrophic Cardiomyopathy (HCM) symptom improvement post mavacamten treatment initiation | Up to 33 months

SECONDARY OUTCOMES:
Participant obstructive Hypertrophic Cardiomyopathy (oHCM) symptoms | Baseline and index date
Participant family history of Hypertrophic Cardiomyopathy (HCM) or obstructive Hypertrophic Cardiomyopathy (oHCM) | Baseline, index date, and up to 33 months
Participant family history of sudden cardiac death (SCD) | Baseline, index date, and up to 33 months
Cardiovascular (CV) and CV-related comorbidities | Baseline
  Including:
  * Aortic stenosis
  * Cardiomyopathies
  * Chronic kidney disease
  * Coronary heart disease
  * Heart failure
  * Hyperlipidemia
  * Hypertension (primary)
  * Hypertensive renal disease
  * Mitral valve prolapse
  * Peripheral vascular disease
  * Pulmonary hypertension
  * Phenocopy disorders (athlete's heart, hypertensive heart disease, Fabry disease, Pompe disease, Danon disease, amyloidosis)
Non-cardiovascular (non-CV) comorbidities | Baseline
  Including:
  * Anxiety/panic attacks
  * Asthma
  * COPD
  * Depression
  * Diabetes
  * Liver disease
Participant electrocardiogram (ECG) rhythm results | Baseline
Participant echocardiogram (ECHO) results | Baseline and index date
Participant cardiac MRI results | Baseline
Participant NT-proBNP results | Baseline
Participant cardiac tropin results | Baseline
Participant cardiopulmonary exercise test (CPET) results | Baseline
Participant cardiac monitoring results | Baseline
Participant exercise test results | Baseline
Hypertrophic Cardiomyopathy (HCM) subtype | Baseline, index date, and up to 33 months
Participant symptoms at Hypertrophic Cardiomyopathy (HCM) | Baseline, index date, and up to 33 months
Participant New York Heart Association (NYHA) class | Baseline, index date, and up to 33 months
Reason/trigger for initiating the path to Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline
Date of reason/trigger that initiated the path to Hypertrophic Cardiomyopathy (HCM) diagnosis | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- IQVIA, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilen O, Adler A, Bastiaenen R, MacNamara JP, Paratz E, Maor E, Arad M, Gold M, Patel N, Pruett C, Burford E, Arora G, Maksabedian Hernandez EJ, Han X, Schuler P, Sandler B, Li L, Tian D, Arora P. Mavacamten Monotherapy in Real-World Patients With Obstructive Hypertrophic Cardiomyopathy: Evidence From COLLIGO-HCM. Circ Genom Precis Med. 2025 Nov 10:e005502. doi: 10.1161/CIRCGEN.125.005502. Online ahead of print. PMID 41212168
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts